CLINICAL TRIAL: NCT06202092
Title: Influence of Honey Phonophoresis on Cartilage Thickness in Patients With Knee Osteoarthritis
Brief Title: Effect of Honey Phonophoresis on Knee Cartilage Thickness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Mohamed Moustafa Mohamed Ahmed, Assistant professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-45/05/851
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Phonophoresis; Ultrasonography

STUDY DESIGN:
Intervention Model Description: Fifty patients with bilateral knee OA whose ages range from 40 to 65 years and body mass indexes between 25 to 35 kg/m2, who will meet the eligibility criteria and will be randomized into two treatment groups using computer-generated numbers in sealed envelopes. The patients will be blinded to the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey Group (Experimental): will receive phonophoresis with honey and conventional physical therapy treatment in the form of transcutaneous electrical nerve stimulation (TENS) current and exercise . The parameters of the application of phonophoresis will be the continuous modality, 1 MHz frequency, intensity of 1 or 1.5 W/cm2, and an application time of 10 minutes
  Interventions: Device: Phonophoresis; Procedure: conventional physiotherapy
- Control Group (Other): will receive ultrasound therapy with gel media and the same conventional physical therapy treatment (control group)
  Interventions: Device: Ultrasound; Procedure: conventional physiotherapy

INTERVENTIONS:
Device: Phonophoresis — Ultrasound using honey as a media over the knee joint
  Arms: Honey Group
Device: Ultrasound — ultrasound using gel as a media over the knee joint
  Arms: Control Group
Procedure: conventional physiotherapy — TENS, Strengthening, and stretching exercises

SUMMARY:
Osteoarthritis (OA) is a progressive chronic disease with the loss of articular cartilage. It is now well recognized that the progression of the disease involves erosion of the cartilage, osteochondral inflammatory damage, and bone distortion. Many recent medical procedures provide treatment through improving symptoms through tissue regeneration and restoring homeostasis to local cells. Unlike bone, articular cartilage is rather recalcitrant to regenerate. Honey is a natural material contain 200 distinct chemical compounds in honey including a wide range of phenolic compounds that have antioxidant, bacteriostatic, antimicrobial, and anti-inflammatory properties. Honey was found to increase the printability and chondrogenic potential of a naturally derived bioink are the main formulations used as hydrogel for Articular Cartilage (AC) regeneration due to their similarity to chondral tissue in terms of morphological and mechanical properties. Design: Double blinded, Randomized control trial. Methods: 50 osteoarthritic patients will be evaluated to be allocated after they match the inclusion criteria then randomized to two groups, group A for Phonophoresis using Honey as coupling media with conventional physical therapy program, group B for ultrasound with regular gel as a coupling media with conventional physical therapy. Outcome measures: the primary outcome measure will be the thickness of the cartilage will be measured using diagnostic ultrasound, the secondary outcome measure will be knee pain measured by the visual analog scale (VAS) and Western Ontario and McMaster Universities OA Index (WOMAC) pain subscale, also functional mobility which will be measured using the stiffness and physical function subscales of the total WOMAC. All will be measured 1 day before starting the procedures and after 4 weeks of the intervention 3sessions/week.

DETAILED DESCRIPTION:
This study will be conducted on patients with bilateral medial tibiofemoral OA, Patients who will be diagnosed and referred by a physician according to the following criteria: bilateral mild-to-moderate medial tibiofemoral OA based on the American College of Rheumatology criteria, and a radiological image (Kellgren-Lawrence Grade II-III). All the patients will be informed about the study and consented to participate in it.

Patients will be excluded from the study if they have rheumatologic conditions such as rheumatoid arthritis, severe knee OA, thrombosis of the lower limbs, physiotherapy treatment of the knee in the previous 6 months, a history of injections in the knee joint during the last 6 months, balance disorders, neuropathy or sensory disorders, skin damage around the knee, previous surgery on the knee joint, or a previous fracture of the lower extremity with knee joint involvement. Patients will be also excluded if they have any contraindications or precautions for the use of ultrasound (e.g., infection, heart problems, pacemaker, metal implants, open epiphysis, pregnancy, thrombophlebitis, or impaired sensation).

Fifty patients with bilateral knee OA whose ages range from 40 to 65 years and body mass indexes between 25 to 35 kg/m2, who will meet the eligibility criteria and will be randomized into two treatment groups using computer-generated numbers in sealed envelopes. The patients will be blinded to the group allocation. Group A will receive phonophoresis with honey and conventional physical therapy treatment in the form of transcutaneous electrical nerve stimulation (TENS) current and exercise (study group). The parameters of the application of phonophoresis will be the continuous modality, 1 MHz frequency, intensity of 1 or 1.5 W/cm2, and an application time of 10 minutes. Group B will receive ultrasound therapy with gel media and the same conventional physical therapy treatment (control group).

Evaluation procedure:

The evaluation process will be conducted within the Department of physical therapy, and Department of radiology of Jazan University, Jazan region, KSA.

The primary outcome measure will be the thickness of the cartilage will be measured using the Versana Essential ultrasound device made in USA using the flat probe 10Hz, the device will measure the cartilage thickness in the middle and posterior medial femoral regions.

The secondary outcome measure will be knee pain measured by the visual analog scale (VAS) and Western Ontario and McMaster Universities OA Index (WOMAC) pain subscale.

The third outcome measure will be functional mobility which will be measured using the stiffness and physical function subscales of the total WOMAC.

Each patient will be assessed 1 day before starting the first session and after the last session according to the same criteria by an assessor who was blinded to the patient's allocation. Initially, all patients will be questioned about their personal data, including age, weight, height, onset and duration of knee pain, and any history of chronic diseases.

Treatment procedure:

The treatment will be conducted in the department of physical therapy, Jazan University, Jazan, KSA.

The total duration of treatment will be 4 weeks, and the treatments will be conducted on alternate days with a frequency of 3 sessions/week. The treatment will target the most affected and painful knee. For patients with equal pain in both knees, the dominant knee was treated. The other knee will take its conventional treatment as an ethical right for the patient to take his/her full treatment.

Both groups will receive the same exercise program during every session for strengthening the quadriceps muscle. The dose will be three sets of ten repetitions, with the starting weight being matched to the ten-repetition maximum weight of each participant. The following quadriceps exercises will be used: (1) quads over a roller (inner range knee extension) using ankle weights for resistance; (2) knee extension in sitting (sitting with the knee at 90° flexion and performing full extension using ankle weights for resistance); (3) straight leg raise (starting in the supine position and raising the leg to 30° hip flexion using ankle weights for resistance); and (4) outer range knee extension (sitting with the knee at 90° flexion and extending to 60° against the resistance of an elastic band). Patients will not be instructed to use any special footwear or insole during treatment to reduce variables and interactions as much as possible.

TENS will be applied to both groups at a frequency of 80 Hz for 20 min (using the Endomed 182 ENRAF NONIUS, Netherlands) through four adhesive electrodes placed over the medial side of the knee region with pulse width constant among all patients and an intensity in the tactile sensation threshold.Ultrasound will be applied to the medial tibiofemoral joint in a continuous mode at a frequency of 1 MHz and an intensity of 1 W/cm2 for a treatment duration of 10 min (Pulson 100 Gymna Uniphy, Belgium) using ultrasound gel for the control group and original honey as a medium under ultrasound head for study group (original honey will be collected from seasonal extracted honey within Jazan region at the time of starting the intervention) for the phonophoresis.

ELIGIBILITY:
Inclusion Criteria:

* bilateral mild-to-moderate medial tibiofemoral Osteoarthritis

Exclusion Criteria:

1. rheumatologic conditions such as:

   * rheumatoid arthritis,
   * severe knee OA,
   * thrombosis of the lower limbs,
2. patients who had physiotherapy treatment of the knee in the previous 6 months,
3. a history of injections in the knee joint during the last 6 months,

   * balance disorders,
   * neuropathy or sensory disorders,
   * skin damage around the knee,
   * previous surgery on the knee joint, or a previous fracture of the lower extremity with knee joint involvement.
4. Patients will be also excluded if they have any contraindications or precautions for the use of ultrasound (e.g., infection, heart problems, pacemaker, metal implants, open epiphysis, pregnancy, thrombophlebitis, or impaired sensation)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
cartilage thickness | 4 weeks
  knee joint cartilage thickness

SECONDARY OUTCOMES:
Pain severity | 4 weeks
  measurment of knee pain using Visual analogue scale which is a straight horizontal line of 100 mm. The ends are defined as the extreme limits of the pain orientated from the left (Best) to the right (Worst).
Functional mobility | 4 weeks
  Using The Western Ontario and McMaster Universities Arthritis Index which is consisting from consisting of 24 items divided into 3 subscales: Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright. Scores range from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status. The higher the score, the poorer the function.

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman Elsayegh, Associate professor, Principal Investigator — University of Jazan
Locations (1):
- Jazan University, Jizan, Gizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No